CLINICAL TRIAL: NCT03642808
Title: Optimisation of Falls Prevention After Low-energy Osteoporotic Fractures: Feasibility Study Based on a Rheumatology-rehabilitation Collaboration
Brief Title: Optimisation of Falls Prevention After Low-energy Osteoporotic Fractures: Feasibility Study
Acronym: OPTICHUTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Hôpital Sainte-Marie Paris (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OPTICHUTE
Record Dates: First submitted 2018-08-08; First posted 2018-08-22 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rehabilitation program (Experimental): * Duration of 8 weeks for a cycle of rehabilitation at the rate of two half-days per week
  * Two interventions per half-day: 30 minutes of education and 1h30 of rehabilitation: physiotherapist, psychomotricity, adapted physical activity
  Interventions: Other: rehabilitation program

INTERVENTIONS:
Other: rehabilitation program — Availibility of patients to complete a rehabilitation program during 8 weeks and to come back 4 times for a careful medical examination

SUMMARY:
Within the Groupe Hospitalier Paris Saint-Joseph (GHPSJ), a reinforced medical care of osteoporosis ('Fracture Liaison service') was organized for osteoporotic fractured patients. The evaluation of benefits of this program through a randomized study showed an improvement in diagnostic tests performed (bone densitometry) and antiosteoporotic treatment initiated (OPTIPOST study, being published in BMJ). However, of 323 patients included, 91 presented a new fracture within 12 months. Among them, 40/126 patients (31.7%) were in the reinforced medical care arm. This result clearly demonstrates the need for a specific medical care program for patients with osteoporotic fracture falling regularly.

DETAILED DESCRIPTION:
Only few studies for secondary prevention of falls have been conducted in France yet. This can be partly explained by the complexity of reeducation programs to implement and by organization issues. Moreover, to our knowledge, no study has demonstrated the benefit of such programs on secondary prevention of osteoporotic fractures, even though falls prevention is needed. Our objective is to demonstrate with a pilot study the feasibility of a falls secondary prevention program, based on a rheumatology (GHPSJ) and reeducation wards (Hôpital Sainte-Marie Paris : HSMP) collaboration. Considering the innovative nature of both this program and this collaboration, a feasibility study is preferable before conducting a larger multicentric study, evaluating locomoter benefits of this program in comparison with usual primary care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (age ≥ 60 years)
* Francophone
* Hospitalized patient or who is consulted in rheumatology or indicated for bone densitometry in Groupe Hospitalier Paris Saint-Joseph, who are suffered a low-energy osteoporotic fracture in the last 12 months
* Patient with an acceptable handicap level definied by a Timed Up & Go test (TUG) <14 seconds
* Autonomous patient with instrumental activities of daily living score (4 items) = 0/4 and Activities of Daily Living score (6 items) ≥5.5/6
* Patient with medical insurance

Exclusion Criteria:

* History of locomor specialized care for the falls prevention
* Cognitive impairment/diagnosed dementia or chronic neurological disorder, which doesn't permit the undertanding or a follow-up to a rehabilitation program
* Fall due to a neurovascular disease or acute cardiovascular
* Significant comorbidities which don't permit a locomotor rehabilitation care
* Refusal to participate in the study
* Refusal to follow the entire rehabilitation program
* Geographic remoteness which doesn't permit the movement to the rehabilitation center
* Contreindicated balneotherapy: incontinence, skin disease or cardiovascular disease
* Patient under guardianship or curatorship
* Patient deprived of liberty

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance and satisfaction of patients with reinforced medical care | 2 months
  compliance and satisfaction of patients with reinforced medical care: compliance questionnaire. Evaluation made for the end of the program of reeducation :
  EVALUATION OF PATIENT ATTENDANCE (2 questions):
  1. How many days did you participate in re-education sessions at the Hôpital Sainte-Marie Paris as part of the OPTICHUTE rehabilitation program?
  2. Have you attended all the proposed rehabilitation sessions? (yes/no)
  EVALUATION OF PATIENT SATISFACTION: possible answer: degree of satisfaction (very satisfied/overall Satisfied/overall dissatisfied/ very dissatisfied)
  A: concerning the initial medical examination and the organization of your appointments : 2 questions B: concerning the progress of the reeducation sessions: 5 questions C: concerning the rehabilitation program more generally: 5 questions D: overall assessment - free comment
Satisfaction of health professionals with reinforced medical care: questionnaire. | 2 months
  Satisfaction of health professionals with reinforced medical care: satisfaction questionnaire. Evaluation made for the end of the program of reeducation Sections A and B and D: Hôpital Sainte-Marie Paris staff, Sections C and D: Groupe Hospitalier Paris Saint Joseph staff 12 questions for the sections A-B-C-D with possible answer: degree of satisfaction (very satisfied/rather satisfied/ rather unhappy/ very dissatisfied)
  A. Regarding the rehabilitation program B. Regarding patients C. Regarding the inclusion visit D: Concerning the link between the rheumatology department of the Groupe Hospitalier Paris Saint Joseph and the hospital day of Rehabilitation of the Hôpital Sainte-Marie Paris
  E: Overall assessment: ree comment

SECONDARY OUTCOMES:
Number of news falls | 1 year
  Number of new falls within the year following the beginning of the program
Number of new osteoporotic fractures | 1 year
  Number of new osteoporotic fractures within the year following the beginning of the program
Number of new hospitalizations | 1 year
  Number of new hospitalizations within the year following the beginning of the program

CONTACTS AND LOCATIONS:
Overall Officials: Agnès PORTIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] McLellan AR, Gallacher SJ, Fraser M, McQuillian C. The fracture liaison service: success of a program for the evaluation and management of patients with osteoporotic fracture. Osteoporos Int. 2003 Dec;14(12):1028-34. doi: 10.1007/s00198-003-1507-z. Epub 2003 Nov 5. PMID 14600804
- [Result] Briot K, Cortet B, Thomas T, Audran M, Blain H, Breuil V, Chapuis L, Chapurlat R, Fardellone P, Feron JM, Gauvain JB, Guggenbuhl P, Kolta S, Lespessailles E, Letombe B, Marcelli C, Orcel P, Seret P, Tremollieres F, Roux C. 2012 update of French guidelines for the pharmacological treatment of postmenopausal osteoporosis. Joint Bone Spine. 2012 May;79(3):304-13. doi: 10.1016/j.jbspin.2012.02.014. Epub 2012 Apr 19. PMID 22521109
- [Result] Campbell AJ, Borrie MJ, Spears GF. Risk factors for falls in a community-based prospective study of people 70 years and older. J Gerontol. 1989 Jul;44(4):M112-7. doi: 10.1093/geronj/44.4.m112. PMID 2738307
- [Result] Karlsson MK, Magnusson H, von Schewelov T, Rosengren BE. Prevention of falls in the elderly--a review. Osteoporos Int. 2013 Mar;24(3):747-62. doi: 10.1007/s00198-012-2256-7. Epub 2013 Jan 8. PMID 23296743
- [Result] Briot K. Fracture Liaison Services. Curr Opin Rheumatol. 2017 Jul;29(4):416-421. doi: 10.1097/BOR.0000000000000401. PMID 28426444
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Result] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Result] Byles JE, Leigh L, Vo K, Forder P, Curryer C. Life space and mental health: a study of older community-dwelling persons in Australia. Aging Ment Health. 2015;19(2):98-106. doi: 10.1080/13607863.2014.917607. Epub 2014 Jun 6. PMID 24903196
- [Result] Ibrahim A, Singh DKA, Shahar S. 'Timed Up and Go' test: Age, gender and cognitive impairment stratified normative values of older adults. PLoS One. 2017 Oct 3;12(10):e0185641. doi: 10.1371/journal.pone.0185641. eCollection 2017. PMID 28972994
- [Result] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204